CLINICAL TRIAL: NCT04156295
Title: Percutaneous Mitral Valve Intervention: Predicting Improvements in Left Ventricular Performance
Acronym: PMVI-PiP
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College Hospital NHS Trust (Other); Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: 248271
Record Dates: First submitted 2019-10-16; First posted 2019-11-07 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Mitral Regurgitation; Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood test will be performed as per routine clinical practice less than 3 months prior to cardiac intervention. Additionally a post procedure follow up blood test will be performed (approximately 3-6 months). Aside from routine blood tests, a small volume of additional blood will be obtained and analysed to test for Troponin T, ST2 and Galectin-3. On completion of testing, blood sample will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the role of cardiac imaging combined with demographic, clinical, and biochemical parameters in predicting outcomes following percutaneous mitral valve intervention in order to facilitate more careful risk stratification, interventional planning and avoidance of high risk futile procedures.The principle objective of this study is to determine if transthoracic echocardiography (TTE) can predict changes in left ventricular (LV) size and function following percutaneous mitral valve intervention (PMVI).

DETAILED DESCRIPTION:
Mitral regurgitation (MR) is one of the most common valvular abnormalities affecting an estimated 5 million worldwide. Within Europe it has been recognised as the second most common valve lesion requiring surgery. By 2030, prevalence is expected to more than double as a consequence of an ageing population. Mitral regurgitation can be caused by a range of aetiologies including degenerative or functional abnormalities. Regardless of the underlying cause, severe MR commonly leads to symptoms of breathlessness and/or arrhythmia, frequently requiring hospital admission secondary to decompensated heart failure. Aside from a reduction in cardiac output secondary to the primary lesion, chronic MR also leads to significant left ventricular remodelling with dilatation and dysfunction of the left ventricle. Left untreated, such a lesion carries an annual mortality of 5%.

Conventional mitral valve surgery is the recognised gold standard therapy for patients with moderate to severe or severe mitral regurgitation, symptoms and LV impairment. However for patients with multiple comorbidities and a high surgical risk, percutaneous mitral valve intervention presents a novel viable therapeutic option.

Percutaneous mitral valve intervention offers an alternative to conventional open heart surgery via a minimally invasive route. One such percutaneous technology is the Mitra-Clip which is deployed and positioned to grasp valve leaflets and create a double orifice. The primary aim is to reduce the degree of mitral regurgitation with additional clinical outcomes focussed on symptom relief, enhanced lifestyle and longevity.

Foundation studies focussed on Mitra-clip have supported the usefulness of percutaneous technology with mainstay papers reporting a reduction in mitral regurgitation with improvement in clinical symptoms and quality of life. When compared to conventional surgery this approach has demonstrated high levels of safety and efficacy. Current research has also acknowledged positive left ventricular (LV) remodelling with improvement in ejection fraction and reduction in LV size as a consequence of percutaneous mitral valve intervention.

Cardiac imaging is crucial in the preoperative, device deployment and post intervention phases of PMVI. TTE, recognised as the mainstay imaging modality in valvular heart disease, allows for both quantitative and qualitative evaluation of mitral regurgitation. Moreover, comprehensive assessment of LV size and function can be performed. More recently, very early myocardial impairment has been demonstrated using a number of sophisticated echocardiographic markers. Additionally, functional testing including exercise stress echocardiography has proven diagnostic relevance when uncovering valvular causes of dyspnoea. Unfortunately the usefulness of both of these echo derived markers in patients with significant mitral regurgitation undergoing PMVI is poorly understood, demonstrating the need for further characterisation of these markers in this cohort.

The aim is to assess the impact of percutaneous mitral valve intervention on markers of LV function and the usefulness of functional testing in predicting changes in LV performance. The investigators propose that cardiac imaging, functional testing and clinical and laboratory data can be used to predict changes in left ventricular size and function following percutaneous mitral valve intervention.

Trial objectives and purpose

The purpose of this study is to assess the role of cardiac imaging combined with demographic, clinical, and biochemical parameters in predicting outcomes following percutaneous mitral valve intervention in order to facilitate more careful risk stratification, interventional planning and avoidance of high risk futile procedures.

The principle objective of this study is to determine if transthoracic echocardiography (TTE) can predict changes in left ventricular (LV) size and function following percutaneous mitral valve intervention (PMVI).

The secondary objectives are:

1. Evaluation of the usefulness of functional testing, namely exercise stress echocardiography (ESE), and its role in discriminating mitral regurgitation (MR) patients who demonstrate improved LV parameters following PMVI from those who do not.
2. Assessment of the relationship between TTE, ESE, Cardiac Magnetic Resonance (CMR) and Cardiac Computed Tomography (CT) for these patients.
3. Assessment of the relationship between improvements in LV performance and the degree of residual MR.
4. Exploration and characterisation of the relationship between changes in LV parameters and clinical outcomes.
5. Assessment of the usefulness of TTE parameters combined with functional, clinical, biochemical parameters in providing a better prediction of postoperative outcomes following PMVI.
6. Exploration of the relationship between improved outcomes and right ventricular (RV) size and function and right ventricular systolic pressures (RVSP).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. At least moderate to severe symptomatic mitral regurgitation
3. Life expectancy greater than 1 year post intervention
4. Able to give informed consent

Exclusion Criteria:

1. Patient not eligible for percutaneous mitral valve intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be performed across two sites, namely Guy's and St Thomas' and King' College Hospitals. Patients will be recruited based on referral to GSTT or KCH, a diagnosis of mitral valve disease and clinical eligibility for percutaneous mitral valve intervention.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in LV size | Within 3-6 months post intervention
  Change in LV size by two dimensional linear dimension (cm)
Change in LV volume (2D) | Within 3-6 months post intervention
  Change in LV volume by Simpson's Biplane method (mL)
Change in LV volume (3D) | Within 3-6 months post intervention
  Change in LV volume by 3D volume method (mL)
Change in LV systolic function (2D EF) | Within 3-6 months post intervention
  Change in LV systolic function by Ejection Fraction by 2D method (%)
Change in LV systolic function (3D EF) | Within 3-6 months post intervention
  Change in LV systolic function by Ejection Fraction by 3D method (%)
Change in LV systolic function (GLS) | Within 3-6 months post intervention
  Change in LV systolic function by Global Longitudinal strain (GLS) by 3D method
Change in LV systolic function (EF1) | Within 3-6 months post intervention
  Change in LV systolic function by First Phase Ejection Fraction (%)

SECONDARY OUTCOMES:
Change in clinical outcomes - symptoms | Within 3-6 months post intervention
  Change in symptoms ( Borg scoring; 0 - lowest = 10 - highest.)
Change in clinical outcomes - NYHA class | Within 3-6 months post intervention
  Change in NHYA class (NHYA class grading)
Change in clinical outcomes - Quality of Life | Within 3-6 months post intervention
  Change in quality of life (Short Form (36) Health Survey) (Score 0-most disability; 100-least disability).
Change in clinical outcomes - 6MWT | Within 3-6 months post intervention
  Change in exercise capacity (6 min walk test distance in metres)
Change in clinical outcomes - NT Pro BNP | Within 3-6 months post intervention
  Change in biomarkers - NT pro BNP (ng/L)
Change in clinical outcomes - ST2, Gal-3, TropT | Within 3-6 months post intervention
  Change in biomarkers - ST2, Galectin 3 and Trop T (ng/mL)
Change in clinical outcomes - residual MR | Within 3-6 months post intervention
  Change in degree of mitral regurgitation (severity grading; 0-none or trivial; 4-severe)
Change in clinical outcomes - RV S' | Within 3-6 months post intervention
  Change in right ventricular performance (RV S' (ms))
Change in clinical outcomes - RV Strain | Within 3-6 months post intervention
  Change in right ventricular performance (strain %)
Change in clinical outcomes - RV Strain Rate | Within 3-6 months post intervention
  Change in right ventricular performance (s-1; (strain per time unit equals velocity difference per unit length).
Change in clinical outcomes - RVSP | Within 3-6 months post intervention
  Change in right ventricular performance (Right ventricular systolic pressure - mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Prendergast, B Med Sc DM, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Given this is a pilot study with much of the data a result of tests considered routine practice, the project is unlikely to generate new IP. However any new IP generated by the research will be owned by Guy's and St Thomas' NHS Foundation Trust. We will not share the data we collect as we have not consented for this however we aim to publish and disseminate our anonymised findings so that the value of this information can be used and applied by others working in the same field.

REFERENCES:
- [Background] Attizzani GF, Fares A, Tam CC, Padaliya B, Mazzurco S, Popovich KL, Davis AC, Staunton E, Bezerra HG, Markowitz A, Simon DI, Costa MA, Sareyyupoglu B. Transapical Mitral Valve Implantation for the Treatment of Severe Native Mitral Valve Stenosis in a Prohibitive Surgical Risk Patient: Importance of Comprehensive Cardiac Computed Tomography Procedural Planning. JACC Cardiovasc Interv. 2015 Sep;8(11):1522-1525. doi: 10.1016/j.jcin.2015.04.025. Epub 2015 Aug 19. No abstract available. PMID 26298225
- [Background] Bonow RO, Carabello BA, Chatterjee K, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2008 focused update incorporated into the ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to revise the 1998 guidelines for the management of patients with valvular heart disease). Endorsed by the Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2008 Sep 23;52(13):e1-142. doi: 10.1016/j.jacc.2008.05.007. No abstract available. PMID 18848134
- [Background] De Backer O, Piazza N, Banai S, Lutter G, Maisano F, Herrmann HC, Franzen OW, Sondergaard L. Percutaneous transcatheter mitral valve replacement: an overview of devices in preclinical and early clinical evaluation. Circ Cardiovasc Interv. 2014 Jun;7(3):400-9. doi: 10.1161/CIRCINTERVENTIONS.114.001607. No abstract available. PMID 24944303
- [Background] Kelley C, Lazkani M, Farah J, Pershad A. Percutaneous mitral valve repair: A new treatment for mitral regurgitation. Indian Heart J. 2016 May-Jun;68(3):399-404. doi: 10.1016/j.ihj.2015.08.025. Epub 2016 Jan 12. PMID 27316505
- [Background] Feldman T, Kar S, Elmariah S, Smart SC, Trento A, Siegel RJ, Apruzzese P, Fail P, Rinaldi MJ, Smalling RW, Hermiller JB, Heimansohn D, Gray WA, Grayburn PA, Mack MJ, Lim DS, Ailawadi G, Herrmann HC, Acker MA, Silvestry FE, Foster E, Wang A, Glower DD, Mauri L; EVEREST II Investigators. Randomized Comparison of Percutaneous Repair and Surgery for Mitral Regurgitation: 5-Year Results of EVEREST II. J Am Coll Cardiol. 2015 Dec 29;66(25):2844-2854. doi: 10.1016/j.jacc.2015.10.018. PMID 26718672
- [Background] Pedrazzini GB, Faletra F, Vassalli G, Demertzis S, Moccetti T. Mitral regurgitation. Swiss Med Wkly. 2010 Jan 23;140(3-4):36-43. doi: 10.4414/smw.2010.12893. PMID 19950042
- [Background] Poulin F, Carasso S, Horlick EM, Rakowski H, Lim KD, Finn H, Feindel CM, Greutmann M, Osten MD, Cusimano RJ, Woo A. Recovery of left ventricular mechanics after transcatheter aortic valve implantation: effects of baseline ventricular function and postprocedural aortic regurgitation. J Am Soc Echocardiogr. 2014 Nov;27(11):1133-42. doi: 10.1016/j.echo.2014.07.001. Epub 2014 Aug 7. PMID 25125314
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698